CLINICAL TRIAL: NCT07091331
Title: Clinical Evaluation of 3D-printed Ceromer Crowns Versus Stainless Steel in Posterior Primary Molars
Brief Title: 3D-printed Ceromer Crowns Versus Stainless Steel in Posterior Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Alan Velazquez, D.D.S., M.P.H., Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2735
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Caries, Dental; Caries; Dentin; Dental Caries in Children
Keywords: Printing, Three-dimensional; Pediatric Dentistry; Tooth, Deciduous; Esthetics, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the esthetic nature of the different materials, masking of the participants and investigators is not possible, however outcomes assessor with be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3D-printed ceromer crown (Experimental): Group A: 3D-printed ceromer crown (Sculpture, Rodin Resins, La Brea, CA, USA)
  Interventions: Procedure: Personalized 3D-printed pediatric ceromer crown
- Stainless steel crown (Active Comparator): Group B: Stainless steel crown (3M Espe, Saint Paul, MN, USA)
  Interventions: Device: Prefabricated stainless steel crown group

INTERVENTIONS:
Procedure: Personalized 3D-printed pediatric ceromer crown — After primary molar crown preparation, digital impression using intraoral scanner (i700, Medit, Seoul, South Korea), crown will be designed with CAD software (CliniCAD, medit, South Korea) and fabricated using a 3D printer, (Sonic mini 4k, Phrozen, Taipei, Taiwan). Crown will be cemented by passive seating using a self-adhesive dual cure cement (Beauticem, shofu, San Marcos, CA, USA)
  Arms: 3D-printed ceromer crown
Device: Prefabricated stainless steel crown group — Stainless steel crown application: After preparation of the tooth, the crown will be filled and cemented with type-1 glass ionomer cement (Ketac Cem easymix, 3M ESPE, Minnesota, USA)
  Arms: Stainless steel crown

SUMMARY:
The aim of the study is to compare preformed metal crowns and 3D-printed ceromer crowns in primary molars of 4-9 years old children. The main questions it aims to answer are:

* How does 3D-printed ceromer crowns compare clincally to stainless steel crowns when restoring posterior molars?
* What is the level of satisfaction of the patient with both materials?
* What is the level of parental satisfaction with both materials?

Study methodology:

This study is a split-mouth clinical trial where participants will receive at least one of each materials in different quadrants of the mouth.

DETAILED DESCRIPTION:
This randomized clinical trial is designed following the Consolidated Standards of Reporting Trials (CONSORT) guidelines and will adopt a prospective, split-mouth approach. The objective is to compare the clinical performance of crowns fabricated with three-dimensional (3D) printed ceromer material against conventional preformed stainless steel crowns in extensively decayed primary posterior teeth. The unit of observation will be gingival inflammation in the area surrounding the restorations, evaluated at specific time points over a 12-month follow-up period (3, 6 and 12 months).

Each eligible participant will receive both types of crowns, with assignments made to contralateral quadrants of the mouth to allow for within-subject comparison. This methodology minimizes inter-individual variability and strengthens internal validity. The ceromer crowns will be fabricated via additive manufacturing (3D printing), while the stainless steel crowns will follow the conventional selection and crimping technique.

Written informed consent will be obtained from their guardians or parents. An expected total of 50 primary molars of healthy participants will be restored.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 9 years with at least 2 primary molars affected by deep occlusoproximal caries.
* Teeth may require pulp therapy (pulpotomy or pulpectomy) and be suitable for full-coverage restoration.
* Teeth must have an antagonist and be located in opposing hemiarches.
* The affected primary molars must be expected to remain in the mouth for at least 12 months.
* The child must be in general good health.
* Parents or legal guardians must sign informed consent, and the child must provide assent.
* Patient does not come to control appointment or does not want to continue research.

Exclusion Criteria:

* Children with systemic diseases or medical conditions affecting oral health.
* Uncooperative behavior (Frankl scale 3 or 4).
* Temporomandibular joint disorders or parafunctional habits (e.g., bruxism).
* Absence of antagonist or adjacent teeth in the selected quadrants.
* Children on long-term medication.
* Patient with allergy to local anesthetic, nickel or chromium.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Plaque index (PI) (Silness and Loe, 1964) | 12 months
  0- No plaque in the area adjacent to the gingiva
  1. There is a thin film on the edge of the gingival margin. (detected with the help of a probe)
  2. There is presence of plaque in the gingival pocket and gingival margin at a level that can be determined by eye. There is no plaque in the proximal area.
  3. A large amount of plaque layer is observed in the gingival pocket and gingival margin. Interdental area is filled with plaque.
Gingival Index (GI) (Loe & Silness, 1963) | 12 months
  0- Healthy gingiva, no inflammation
  1. Mild inflammation, discoloration and mild edema of the gums, no bleeding on probing.
  2. Moderate inflammation, redness and edema in gums, bleeding on probing.
  3. Advanced inflammation, redness, edema in gums, spontaneous bleeding is observed.
International Dental Federation (FDI) criteria used for clinical evaluation of indirect restorations | 12 months
  Functional, Biological and Esthetic properties, scored from 1-5 (higher score meaning worse result.

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  A 5 question satisfaction questionnaire with 5 point lykert scale questions
Parental satisfaction | 6 months
  A 5 question satisfaction questionnaire with 5 point lykert scale questions

CONTACTS AND LOCATIONS:
Overall Officials: Alan Velazquez, DDS, MPH, Principal Investigator — Universidad Autonoma de Baja California
Locations (1):
- Facultad de Odontología, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared to with